CLINICAL TRIAL: NCT03533816
Title: Phase I Study of Ex Vivo Expanded/Activated Gamma Delta T-cell Infusion Following Haploidentical Hematopoietic Stem Cell Transplantation and Post-transplant Cyclophosphamide
Brief Title: Expanded/Activated Gamma Delta T-cell Infusion Following Hematopoietic Stem Cell Transplantation and Post-transplant Cyclophosphamide
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: In8bio Inc. (Industry)
Responsible Party: Principal Investigator, Joseph McGuirk, Professor & Division Director, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-Gamma-DeltaTcell
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes
Keywords: Gamma delta T-cells; Hematopoietic Stem Cell Transplantation (HCT); Post-transplant Cyclophosphamide (PTCy); Expanded/Activated gamma delta (EAGD); Graft versus host disease (GVHD); haploidentical
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Graft vs Host Disease | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Intervention Model Description: This dose escalation study will be conducted in two phases. The first phase will have three cohorts with three recipient/donor pairs at different dose levels for each cohort. The second phase is an expansion cohort at the maximum tolerated dose determined in the first phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EAGD T-cell infusion (Phase I) (Experimental): Peripheral blood is collected by leukapheresis from the donor, expanded and activated on CliniMACS-Prodigy, further depleted of alpha beta T-cells using the CliniMACS Alpha Beta T-Cell Depletion System, which leaves a gamma delta T-cell rich product. This product is then infused into the recipient at either 1, 3, or 10 x 1,000,000 cells/kg concentrations depending upon the cohort.
  Interventions: Drug: EAGD T-cell infusion (Phase I)
- EAGD T-cell infusion (Expansion) (Experimental): Peripheral blood is collected by leukapheresis from the donor, expanded and activated on CliniMACS-Prodigy, further depleted of alpha beta T-cells using the CliniMACS Alpha Beta T-Cell Depletion System, which leaves a gamma delta T-cell rich product. This product is then infused into the recipient at the maximum tolerated dose as determined from Phase I.
  Interventions: Drug: EAGD T-cell infusion (Expansion)

INTERVENTIONS:
Drug: EAGD T-cell infusion (Phase I) — The Alpha Beta (α/β) T-Cell Depletion System utilizes the CliniMACS instrument to yield a gamma delta (γδ) enriched cell therapy product.
  Other Names: CliniMACS-Prodigy; CliniMACS Alpha Beta T-Cell Depletion System
  Arms: EAGD T-cell infusion (Phase I)
Drug: EAGD T-cell infusion (Expansion) — The Alpha Beta (α/β) T-Cell Depletion System utilizes the CliniMACS instrument to yield a gamma delta (γδ) enriched cell therapy product.
  Other Names: CliniMACS-Prodigy; CliniMACS Alpha Beta T-Cell Depletion System
  Arms: EAGD T-cell infusion (Expansion)

SUMMARY:
Gamma delta T-cells are part of the innate immune system with the ability to recognize malignant cells and kill them. This study uses gamma delta T-cells to maximize the anti-tumor response and minimize graft versus host disease (GVHD) in leukemic and myelodysplastic patients who have had a partially mismatched bone marrow transplant (haploidentical).

DETAILED DESCRIPTION:
Many patients with hematological malignancies require a bone marrow transplant for curative treatment. A matched sibling donor is optimal but may not be available. Therefore, a partially matched family member (haploidentical) may be a viable alternative. The incidence of graft vs. host disease, however, can become more of a significant, even fatal, factor with partial matches.

T-cells have been shown to be the key player in the post-transplant immune phenomena. The majority of T-cells are composed of alpha beta T-cells with a small minority of gamma delta T-cells, which are known to have the unique ability to kill malignant cells without antigen recognition.

This study proposes to extract, concentrate, and activate gamma delta T-cells from the peripheral blood to provide innate anti-tumor effect with minimal risk of GVHD. Safety and impact and/or the rate of GVHD will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

The following criteria are used to enroll patients in the study before transplant.

* Patients with neoplastic hematological disorders with indication of allogeneic transplant according to the National Comprehensive Cancer Network (NCCN) or other standard guidelines as follows:

  * Acute myeloid leukemia [AML] in morphologic complete remission with intermediate/high-risk features (per NCCN criteria) or relapsed disease
  * Chronic myeloid leukemia [CML] in any chronic phase.
  * Myelodysplastic syndrome [MDS] with intermediate/high risk features or refractory disease (with bone marrow blast count <10%).
  * Acute lymphoblastic leukemia [ALL] in morphologic complete remission with high-risk features or relapsed disease.
* Negative test for donor-specific antibody within 28 days of starting conditioning regimen.
* Age Criteria: 19-65 years.
* Organ Function Criteria: The following organ function testing should be done within 35 days before study registration.

  * Cardiac: Normal left ventricular ejection fraction (LVEF) (50% or above) as measured by MUGA or Echocardiogram.
  * Pulmonary: FVC, FEV1 and DLCO (corrected) should be 50% or above of expected.
  * Renal: serum creatinine level to be <2 mg/dl AND estimated (Cockcroft-Gault formula) or measured (takes priority if done) creatinine clearance (CrCl) must be equal or greater than 70 mL/min/1.73 m2.
  * Hepatic: serum bilirubin 1.5 upper limit of normal (ULN), Aspartate transaminase (AST)/alanine transaminase (ALT) 2.5 ULN, and alkaline phosphatase 2.5 ULN.
* Performance status: Karnofsky performance score (KPS) or Lansky score: ≥80.
* Hematopoietic cell transplant comorbidity index (HCT-CI) <3. Exception may be made on individual cases after discussion with the primary investigator.
* Consent: All patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.

The following criteria are required within 48 hours prior to infusion of the EAGD T cell product.

* Absence of uncontrolled infection with sepsis syndrome (e.g persistent positive blood culture).
* NO hemodynamic instability (due to sepsis or organ dysfunction) or circulatory volume overload.
* NO clinically significant organ toxicity that are defined as follows:

  * Heart failure with subnormal LVEF or clinical fluid overload.
  * Elevated serum creatinine or subnormal creatinine clearance (either estimated or measured).
  * Elevated total bilirubin ≥1.5 upper normal level (unless indirect hyperbilirubinemia attributed to non-hepatic pathology), or elevated liver enzymes (ALT, AST, ALP) >5 x ULN.
  * Hypoxemia requiring oxygen therapy
* NO acute graft versus host disease (any grade).
* Neutrophil engraftment.

Exclusion Criteria:

* Non-compliant patients.
* No appropriate caregivers identified.
* Uncontrolled medical or psychiatric disorders which may preclude patients to undergo clinical studies (Discretion of the attending physician).
* Active central nervous system (CNS) neoplastic involvement.
* Morbid obesity with body mass index >35 (borderline cases may be considered on case-by-case basis after discussion with the primary investigator).
* Patients with known allergy to DMSO.
* HIV1 (Human Immunodeficiency Virus-1) or HIV2 positive.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Phase I - Dose-limiting toxicity (DLT) | Baseline to Day 30
  The dose escalation strategy will follow the Food and Drug Administration Guideline for design of early phase clinical trials of cellular therapy products.
Phase I - Severe acute adverse events following infusion of EAGD T-cells | Baseline to Day 100
  Safety of the infusion will be based on the risk of treatment-related severe adverse events as identified in the National Cancer Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Expansion phase - Rate of acute GVHD | Baseline to Day 100
  Monitoring for GVHD is assessed with Grade II-IV adverse events as identified by the National Cancer Common Terminology Criteria for Adverse Events (CTCAE) version 4.

SECONDARY OUTCOMES:
Expansion phase - Relapse following haploidentical HCT and PTCy with EAGD T-cell infusion | Baseline to 100 days
  Number of subjects who have acute GVHD by day 100 post-HCT after infusion of EAGD T-cells
Expansion phase - Non-relapse mortality following haploidentical HCT and PTCy with EAGD T-cell infusion | Baseline to 100 days
  Number of subjects who have no relapse by day 100 post-HCT after infusion
Expansion phase - Overall survival following haploidentical HCT and PTCy with EAGD T-cell infusion | Baseline to 100 days
  Number of subjects who are living by day 100 post-HCT after infusion
Rate of one-year relapse-free survival (RFS) | Baseline to one year
  Number of subjects living without relapse of disease after one year following HCT
Rate of one-year non-relapse mortality (NRM) | Baseline to one year
  Number of subjects no longer living but not from disease relapse after one year following HCT
Rate of one-year overall survival (OS) | Baseline to one year
  Number of subjects living after one year following HCT
Proportion of subjects with chronic GVHD at one year | Baseline to one year
  Number of subjects with chronic GVHD after one year following HCT

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McGuirk, M.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Cancer Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No